CLINICAL TRIAL: NCT06201221
Title: Advantages of Single-port Laparoscopy in the Treatment of Benign Ovarian Tumors in Children and Adolescents: A Multicenter Retrospective Study
Brief Title: Single-port Laparoscopy in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Collaborators: Quanzhou First Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Yebin Feng, Director, Fujian Maternity and Child Health Hospital
Other Study IDs: FujianMCHH-Tong01
Record Dates: First submitted 2023-12-09; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Benign Ovarian Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single-port Laparoscopy group: Single-port Laparoscopy in the Treatment of Benign Ovarian Tumors in Children and Adolescents
  Interventions: Procedure: single-port laparoscopy surgery
- Multiport Laparoscopy group: Multiport Laparoscopy in the Treatment of Benign Ovarian Tumors in Children and Adolescents
  Interventions: Procedure: multiport laparoscopy surgery

INTERVENTIONS:
Procedure: single-port laparoscopy surgery — The two groups underwent different surgical procedures.
  Groups: Single-port Laparoscopy group
Procedure: multiport laparoscopy surgery — The two groups underwent different surgical procedures.
  Groups: Multiport Laparoscopy group

SUMMARY:
To compare the safety evaluation, efficacy evaluation, long-term aesthetics and psychological satisfaction of single-port and multiport laparoscopy for children and adolescents with BOT in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤18 years old
* Postoperative pathological diagnosis confirmed benign ovarian tumor
* Multi-hole laparoscopic or single-hole laparoscopic surgery
* Medical records and pathological data were complete and available

Exclusion Criteria:

* Patients with malignant pathological diagnosis
* Patients undergoing open surgery
* Incomplete medical records or pathological data

Ages: 1 Year to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients aged ≤18 years and pathologically diagnosed with BOT were collected from the electronic medical records of six gynecological oncology medical centers in Fujian, China between January 2019 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Operation duration | 3 hours
  The time elapsed from the initial incision to final skin closure

SECONDARY OUTCOMES:
The Visual Analog Scale (VAS) score | 24 hours after surgery
  Postoperative pain was evaluated by The Visual Analog Scale (VAS) score. The scale has a maximum score of 10 and a minimum score of 0, with higher scores meaning worse outcomes
5-point Likert scale | 1 month and 1 year after surgery
  5-point Likert scale to assess the satisfaction at 1 month and 1 year post-operatively. The scale has a maximum score of 5 and a minimum score of 1, with higher scores meaning better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, Ph.D, Principal Investigator — Fujian Maternity and Child Health Hospital
Locations (1):
- Fujian Maternal and Child Health Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT06201221/Prot_000.pdf